CLINICAL TRIAL: NCT03502954
Title: A Phase 1, First-in-human, Randomized, Double Blind, Placebo Controlled, Safety, Tolerability and Pharmacokinetic Study of ABY 039 in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of ABY-039
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Halted prematurely
Sponsor: Affibody (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ABY-039-001; 2017-002918-32 (EudraCT Number)
Record Dates: First submitted 2018-03-23; First posted 2018-04-19 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ABY-039 IV (Experimental)
  Interventions: Biological: ABY-039
- ABY-039 SC (Experimental)
  Interventions: Biological: ABY-039
- Placebo IV (Placebo Comparator)
  Interventions: Biological: Placebo
- Placebo SC (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ABY-039 — ABY-039
  Arms: ABY-039 IV; ABY-039 SC
Biological: Placebo — Placebo
  Arms: Placebo IV; Placebo SC

SUMMARY:
The purpose of this first-in-human study is to investigate the safety and tolerability of ABY-039 after single and multiple doses in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects between 18 to 55 years of age agreeing to use highly effective methods of contraception
2. Body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive, with a weight of at least 50 kg
3. Non-smoker
4. Subjects in good health
5. Subjects with total immunoglobulin G (IgG) > 10 g/L at Screening

Exclusion Criteria:

1. Subjects who have donated blood in the 3 months prior to Screening, plasma in the 7 days prior to Screening or platelets in the 6 weeks prior to Screening
2. Subjects who have received systemic corticosteroid treatment within 3 months of first dosing
3. Subjects who have a history of significant drug allergy (e.g., anaphylaxis) or any clinically significant allergic condition (excluding non-active hay fever), as determined by the investigator
4. Subjects who are still participating in another clinical study or received last investigational medical product (IMP) dose in a clinical study within the following time period prior to dosing: 3 months or 5 half-lives, whichever is longer
5. History of splenectomy, asthma (exception of resolved childhood asthma), or chronic obstructive pulmonary disease (COPD)
6. Positive for hepatitis A, hepatitis B, hepatitis C virus or antibodies to HIV-1 and/or HIV-2 or a positive QuantiFERON Gold Plus test at Screening
7. Subjects who have received a live vaccination within 3 months prior to Screening or plan to have a live vaccination within 3 months after the last dose of study drug
8. Subject unable or unwilling to comply with the protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Number of (related) treatment emergent adverse events of single intravenous (IV) and subcutaneous (SC) infusions/injections, and multiple SC injections | Baseline up-to 11 weeks post-dose
  Determining the incidence, severity, and dose relationship of adverse events that are related to treatment with ABY-039

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MD, Principal Investigator — Parexel
Locations (1):
- PAREXEL Early Phase Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No